CLINICAL TRIAL: NCT03478995
Title: A Phase 1b, Open Label, Dose-escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GX-I7 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Study to Evaluate Safety and Tolerability of GX-I7 in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GX-I7-CA-003
Record Dates: First submitted 2018-01-31; First posted 2018-03-27 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Locally Advanced or Metastatic Solid Tumors
Keywords: Phase1b
MeSH Terms: interventions — efineptakin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GX-I7 (Experimental): Determined dose of GX-I7 on Day1 of each cycle
  Interventions: Drug: GX-I7

INTERVENTIONS:
Drug: GX-I7 — GX-I7 25mg/ml/vial

SUMMARY:
Patients will be enrolled in two stages:

* Dose-escalation stage: Approximately 15-30 patients will be enrolled.
* Dose-expansion stage: 6-12 patients will be enrolled. Dose-escalation slots will be filled first, then dose-expansion slots.

DETAILED DESCRIPTION:
* Dose-escalation stage : designed as classical 3+3 to determine MTD or RP2D to evaluate approximately GX-I7.
* Dose-expansion stage : designed to enroll additional 6-12 patients to acquire additional safety and pharmacodynamic data to more fully inform the dose selection for RP2D

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (ICF)
* Age ≥ 19 years
* Able to comply with the study protocol, in the investigator's judgment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy ≥ 12 weeks
* Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment (Cycle 1, Day 1)
* Serum pregnancy test for women of childbearing potential (including women who have had a tubal ligation) must be performed and documented as negative within 14 days prior to Cycle 1, Day 1
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm
* Patients with histologic documentation of locally advanced, recurrent, or metastatic incurable solid tumors that has progressed after at least one available standard therapy; or for whom standard therapy has proven to be ineffective or intolerable, or is considered inappropriate
* Patients with measurable disease per RECIST v1.1

Exclusion Criteria:

* Inability to comply with study and follow-up procedures
* Pregnancy, lactation, or breastfeeding
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 3 months, unstable arrhythmias, and/or unstable angina
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, and inherited liver disease or current alcohol abuse
* Poorly controlled Type 2 diabetes mellitus defined as a screening hemoglobin A1C ≥ 8% or a fasting plasma glucose ≥ 160 mg/dL (or 8.8 mmol/L)
* Major surgical procedure within 28 days prior to Cycle 1, Day 1, or anticipation of need for a major surgical procedure during the study
* Any anti-cancer therapy, whether investigational or approved, including chemotherapy, hormonal therapy, and/or radiotherapy, within 3 weeks prior to initiation of study treatment
* Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤ 1 except for alopecia, vitiligo, or endocrinopathy managed with replacement therapy
* History of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
* Primary CNS malignancy, untreated CNS metastases, or active CNS metastases (progressing or requiring corticosteroids for symptomatic control)
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
DLT | up to 24 months
  Incidence of nature of DLTs
AE | up to 24 months
  Incidence, nature and severity of adverse events graded according to NCI CTCAEv4.0
ECG test evaluated by QTc | up to 24 months
  Change QTc from baseline (> 500 msec)

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile | up to cycle 3 day 1(approximately 9 weeks)
  Serum concentration of GX-I7 at specified timepoints for the Area under the concentration time-curve (AUC)
Anti-tumor activity | up to 24 months
  Objective response, defined as a complete response (CR) or partial response (PR) per RECIST v.1.1, as determined by the investigator
Immunogenicity | up to 24 months
  Incidence of anti-drug antibodies (ADAs) during the study
Exploratory Biomarker | up to 24 months
  Changes in immune infiltrates, immune-related gene expression in tumor tissue prior to and during study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joo Hyuk Sohn, MD, Principal Investigator — Yonsei University Health System, Severance Hospital; Tae Won Kim, MD, Principal Investigator — Medical Oncology, Asan Medical Center; Myoung-Ah Lee, MD, Principal Investigator — Medical Oncology, Seoul St. Mary's Hospital, of the Catholic University
Locations (3):
- South Korea (3):
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Seoul St. Mary's Hospital, of the Catholic University, Seoul

REFERENCES:
- [Derived] Kim GM, Kim S, Lee MA, Byun MS, Choi D, Yang SH, Woo J, Sung YC, Shin EC, Park SH, Kim TW, Sohn J. GX-I7, a long-acting IL-7, safely and effectively increased peripheral CD8+/CD4+ T cells and TILs in patients with locally advanced or metastatic solid tumours. Br J Cancer. 2025 Sep;133(4):524-532. doi: 10.1038/s41416-025-03069-3. Epub 2025 Jun 9. PMID 40490502